CLINICAL TRIAL: NCT03095430
Title: Modulation of General Anesthesia Using Entropy and Surgical Pleth Index
Acronym: ESPTR
Status: Completed | Type: Observational
Sponsor: Romanian Society of Anesthesia and Intensive Care (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Alexandru Florin Rogobete, Principal Investigator, Romanian Society of Anesthesia and Intensive Care
Other Study IDs: 20161213CA
Record Dates: First submitted 2017-03-07; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Trauma; General Anaesthetic Drug Overdose
Keywords: Trauma; General Anesthesia; Surgical Pleth Index; Entropy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPI Group: General Anesthesia using Entropy and Surgical Pleth Index Monitoring
  Interventions: Device: Monitoring
- Control Group: General Anesthesia without Entropy and Surgical Pleth Index (Control Group)

INTERVENTIONS:
Device: Monitoring — Monitoring
  Groups: ESPI Group

SUMMARY:
The critically ill polytrauma patient is one of the most complex cases with regard to the optimization of the intensive care, anesthesia, as well as postoperative management. One of the most important steps in the complex management of such patients is the modulation of anesthesia and the volemic resuscitation, especially in the first hours post-trauma, and in the operating room admission. We start with the assumptions that the optimization of anesthesia should depend on each patient, being conducted in an individual manner. We also believe that by individualizing the anesthesia by monitoring the entropy and SPI it is possible to obtain an appropriate management regarding resuscitation and volume replacement. Furthermore it assumes that an adequate anesthesia, and resuscitation singled volume replacement can reduce morbidity and mortality rates as well as the period of stay in the ICU and recovery time.

DETAILED DESCRIPTION:
Objectives

The project aims to aid to the Romanian healthcare system, by assuring new modernized monitoring equipment, specific for the department of anaesthesia and intensive care, for both clinical and paraclinical data, as well as for the existing information for modulation and optimizing of the general anaesthesia used in critically ill polytrauma cases based on modern techniques, such as entropy, and surgical pleth index (SPI). In this way, it aims to create a new prospect of developing a model, which will help the physicians in the decision-making process, hoping to improve the stats in the high morbidity and mortality rates in this specific field of medicine.

Reducing the mortality and increasing the quality of the provided medical services is possible by assuring a modern monitoring system, because critically ill patients should be observed through complex techniques. Furthermore, interpretation and timely synthesis of the biological signals and their correlation with other clinical and laboratory data are useful in modulating general anesthesia in the critically conditions.

General objectives comprise of developing a new research field regarding the international standards of research and combating the economic and social needs of Romania and Europe, by creating a complete protocol, which is innovative and helpful in improving the mortality and morbidity index for polytrauma patients admitted in the intensive care unit (ICU), by means of better monitoring procedures and modulating the anaesthesia and therapeutic management, therefore increasing the efficiency of the public health care system.

The specific objectives of the study are to represent the integration of modern anesthesia methods used for monitoring and optimizing the management of anesthesia and therapy options, depending on each patient as an individual; calculating the severity scores and risk factors, both in the first 24 hours as well as continuously, providing support instruments designed to add to the medical decision making process, and make it possible in a very short time, developing an ergonomic mode, dynamic and standardized viewing of local and distant perioperative anesthetic protocols, modulated by non-invasive modern techniques for anaesthesia monitoring.

Measurements:

All the patients enrolled in the study will have a monitoring sheet from the start, which will contain details regarding the following: a) Demographic data: age, sex, BMI (registered at the time of admission); b) Clinical data: ASA score, ISS score, APACHE II score, trauma mechanism, type of surgical intervention (registered at the time of admission); c) Laboratory data: EAB parameters, complete blood count, fibrinogen, ESR, PCR, total bilirubin (T0 - before orotracheal intubation, T1 - at extubating, T2 - at 24 hours post-operatively, T0 - before orotracheal intubation, T2 - at 24 hours post-operatively; d) Clinical parameters: heart rate, mean blood pressure, SpO2 plethysmography, EtCO2 capnography, entropy, SPI, axillary skin temperature probe, diuresis (T0 - before orotracheal intubation, at an interval of 15 minutes perioperative, T1 - at extubating); e) Perioperative events: hypotension, bradycardia, bronchospams, SpO2 drop (desaturation) lower than 90% via pulse oximetry (Every event should be noted in the monitoring sheet of the study); f) Events related to intubation: laryngospasms, failed intubation, tissue injury resulting from difficult intubating conditions, postoperative airway complications due to difficult intubation (Every event should be noted in the monitoring sheet of the study). The database officer should register all the patient data relevant for the study in electronic format including all details noted in the monitoring sheet.

Statistical Analysis:

For statistically analysis of the study, in concordance to these objectives, a series of statistical tests were utilized which can satisfy all the statistical objectives of the study. For analysis if the normal distributions of continuous data, the Kolmogorov-Smirnov test will be utilized. Similarly, data with a normal distribution were compared using the Student t test and presented as mean with SD. Last but not the least, data with an inhomogeneous distribution will be compared using the Mann-Whitney U test and presented as median. Nominal data will be compared using the chi-square test. For highlighting the statistical differences, a P value less than 0.05 was considered as significant. The statistical analysis of data will be performed computerized with the programs Microsoft Office Excel for Mac 2011 v.14.4.7. (Microsoft Corporation, Bucharest, Romania) and Prism 6 for Mac OS X v.6.0. (GraphPad Software, Inc., San Diego, CA). This analysis consisted, in the calculation of frequencies and the percentages for qualitative variables, as well as the calculation of the arithmetic means and the standard deviations for quantitative variables. The statistical estimation of the results was performed using the criteria decision of the statistical test. Similarly, the lot will be further statistically analyzed for determining the heterogeneity/homogeneity in between the groups. Similarly, for increasing in the transparency between the different groups, patients will be divided into more groups, as presented in this study.

ELIGIBILITY:
Inclusion Criteria:

* age limit: between 18 years to 80 years;
* gender: male and female;
* within 2 hours of surgical intervention;
* ASA physical status I, II, III;
* written consent accepted to be enrolled in the study; in polytrauma patients in the operation theatre who are brought directly through the emergency department, written consent is obtained from the relatives, in accordance to the national law number 206, of 2004, for a good and correct scientific research, in the situation where the patient is no capable to sign or give the written consent;

Exclusion Criteria:

* cardiac pacemaker;
* atrial fibrillation at the time of presentation in the operation theatre;
* any subject with epidural catheter, placed pre-operatively;
* allergy to Propofol or another anesthetic drugs;
* pregnancy;
* presence of neuromuscular disease;
* presence of neurologic disease;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Polytrauma patients admitted in OR
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Change of systolic blood pressure baseline | Change from Baseline Systolic Blood Pressure at 1 hour
  Evaluating the impact of general anesthesia guided with Entropy and SPI on the hemodynamic instability in the critically ill polytrauma patient; hemodynamic instability is represented and characterized by high blood pressure episodes (hypertension), or low blood pressure (hypotension).
Change of heart beat rate baseline | Change from Baseline heart beat rate at 1 hour
  Evaluating the impact of general anesthesia guided with Entropy and SPI on the heart rate in the critically ill polytrauma patient; cardiac rate instability is represented and characterized by high cardiac rate (tachycardia), or low cardiac rate (bradycardia)
Opioid consumption | Through study completion, an average of 1 year
  Evaluating the opioid consumption by general anesthesia-guided with Entropy and SPI

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Rogobete, MSc, PhDs, Clin Res, Principal Investigator — Romanian Society of Anesthesia and Intensive Care; Ovidiu Horea Bedreag, MD, PhD, Asssit Prof, Study Director — Victor Babes University of Medicine and Pharmacy Timisoara; Dorel Sandesc, MD, PhD, Prof, Study Chair — Victor Babes University of Medicine and Pharmacy Timisoara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogobete AF, Sandesc D, Cradigati CA, Sarandan M, Papurica M, Popovici SE, Vernic C, Bedreag OH. Implications of Entropy and Surgical Pleth Index-guided general anaesthesia on clinical outcomes in critically ill polytrauma patients. A prospective observational non-randomized single centre study. J Clin Monit Comput. 2018 Aug;32(4):771-778. doi: 10.1007/s10877-017-0059-2. Epub 2017 Aug 30. PMID 28856631 (Retraction: PMID 31641919 J Clin Monit Comput. 2020 Jun;34(3):619)